CLINICAL TRIAL: NCT02689661
Title: The Impact of the Metabolic Syndrome on the Incidence of Neuropathy in Obese Subjects
Brief Title: Impact of the Metabolic Syndrome on the Incidence of Neuropathy in Obese Subjects
Status: Completed | Type: Observational
Sponsor: Brian Callaghan (Other)
Responsible Party: Sponsor-Investigator, Brian Callaghan, Assistant Professor of Neurology, University of Michigan
Organization: University of Michigan (Other)
Other Study IDs: NINDS-NS079417
Record Dates: First submitted 2016-01-14; First posted 2016-02-24 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Metabolic Syndrome; Obesity; Neuropathy
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma or serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese participants: Obese participants recruited from the University of Michigan Investigational Weight Management Clinic. Subjects in this group complete the five surveys, undergo extensive metabolic phenotyping, and a comprehensive neuropathy assessment at study entry and again at 2 years.
- Lean participants: Healthy lean age and gender matched controls recruited via the umclinicaltrials.org complete the five surveys, complete an oral glucose tolerance test and cholesterol panel, as well as the complete comprehensive neuropathy assessment.

SUMMARY:
The primary purpose of this study is to discover modifiable risk factors for the development of neuropathy, specifically looking at the metabolic syndrome.

DETAILED DESCRIPTION:
The investigators propose to follow obese individuals and determine the impact of the aspects of the metabolic syndrome on the incidence of neuropathy compared to lean individuals.

While there are many well established relationships between obesity and disease, the association of obesity and the metabolic syndrome with peripheral neuropathy is less clear.

The investigators will be following a population of 300 adult individuals age 18 years or older with obesity and 300 adult individuals without obesity or any aspect of the metabolic syndrome (hyperlipidemia, hypertriglyceridemia, hypertension, hyperglycemia, obesity). Obese subjects will be recruited through the Investigational Weight Management Clinic. A proportion of the subjects will be recruited through Blue Care Network of Michigan (BCN) as part of their Healthy Blue Living campaign which is supporting clinical care of up to 400 individuals in the clinic. The individuals not recruited directly through the clinic will be identified via flyer, word of mouth, and umclinicalstudies.org.

The phenotyping information for the obese subjects will be already completed as part of the initial project. Lean subjects will undergo screening for eligibility, which includes taking height, weight, blood pressure, lipid profile, and glucose tolerance test.

Neuropathy measures completed at baseline and 2 years (obese subjects only) include: definite clinical neuropathy will be established using Toronto consensus guidelines based upon neurologic exam, nerve conduction studies, Michigan Neuropathy-Specific Instrument, Utah Early Neuropathy Scale, balance and hip strength measures, cognitive testing (computerized cognitive screening to determine how obesity affects the central nervous system) (also done at time 12 +/- 4 weeks and 52 +/- 4 weeks post-baseline visit), neurothesiometer testing, skin biopsy to determine nerve fiber density, Quantitative Sudomotor Axon Reflex Test (QSART) to measures the autonomic nerves that control sweating, heart rate variability/cardiac autonomic neuropathy testing to assess for autonomic neuropathy, quantitative sensory testing to assess for small fiber neuropathy, Sudoscan to assess sweat gland function, and the following questionnaires: Neuropathy Quality of Life, McGill Pain, Autonomic symptoms profile.

The investigators intend to demonstrate that obesity and other aspects of the metabolic syndrome have a direct impact on the incidence of peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18
2. Willing and able to provide written informed consent, enrolled in the Investigational Weight Management Clinic at the University of Michigan

Exclusion Criteria:

1. Taking blood thinning medications, except aspirin, Evidence of inherited disorders of lipid metabolism
2. History of cancer within the last 5 years
3. Human immunodeficiency virus (HIV) antibody positive
4. Subjects with solid organ transplants
5. Participation in any other clinical trial within 90 days of entry into this trial
6. Pregnant or lactating females
7. Uncontrolled thyroid disease
8. Unstable angina or New York heart association class II failure or above
9. Gastrointestinal disease specifically gastrointestinal motility disorders
10. Unstable neuropsychiatric disease including major depression/anxiety, bulimia, or anorexia
11. End stage renal or hepatic disease
12. Autoimmune disorders (e.g. lupus)
13. Body weight fluctuation of more than 5 kg in the previous 3 months
14. Prior bariatric surgery
15. A history or current substance abuse, change in smoking habits, or cessation in the past 6 months
16. Women of childbearing age must use a reliable form of contraception
17. Any medical condition, which would make the patient unsuitable for recruitment, or could interfere with the patient participating in or completing the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include eligible patients who are currently enrolled in the University of Michigan Investigational Weight Management Clinic as well as age and gender matched lean controls.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2010-11; Primary Completion 2019-07 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Neurologist history and examination for presence of neuropathic symptoms, abnormal sensory examination findings, and abnormal reflexes (no specific instrument) | Baseline
  Toronto definition of probable clinical neuropathy (2 or 3 out of 3 of the following: neuropathic symptoms, sensory examination findings, and reflexes)
Nerve fiber density at the leg | Change from baseline to year 2

SECONDARY OUTCOMES:
Sural sensory nerve conduction amplitude | Baseline and 2 year
  Physiologic parameter
Peroneal motor nerve conduction amplitude | Baseline and 2 year
  Physiologic parameter
Tibial motor nerve conduction amplitude | Baseline and 2 year
  Physiologic parameter

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Callaghan, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Callaghan BC, Xia R, Reynolds E, Banerjee M, Rothberg AE, Burant CF, Villegas-Umana E, Pop-Busui R, Feldman EL. Association Between Metabolic Syndrome Components and Polyneuropathy in an Obese Population. JAMA Neurol. 2016 Dec 1;73(12):1468-1476. doi: 10.1001/jamaneurol.2016.3745. PMID 27802497

DOCUMENTS (1):
  • Informed Consent Form (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT02689661/ICF_000.pdf